CLINICAL TRIAL: NCT06186583
Title: A Mass Balance Study of [14C]ABSK021 in Healthy Adult Male Chinese Subjects
Brief Title: A Mass Balance Study of [14C]ABSK021
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK021-104
Record Dates: First submitted 2023-11-20; First posted 2024-01-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: On Day 1, subjects will receive a single oral dose of approximately 50 mg ABSK021 containing approximately 100 μCi of [14C] ABSK021 in the fasted state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]ABSK021 Suspension (Experimental): On Day 1, subjects will receive a single oral dose of approximately 50 mg ABSK021 containing approximately 100 μCi of [14C] ABSK021 in the fasted state.
  Interventions: Drug: Pimicotinib（ABSK021）

INTERVENTIONS:
Drug: Pimicotinib（ABSK021） — A standard meal should be given to the subjects in the evening before dosing. Then, the subjects should fast for at least 10 hours. Water is not prohibited overnight. The next morning, the subjects should administer study drug in fasted state with warm water. The total volume of warm water and suspension is approximately 240 mL. Water is prohibited from 1 hour before dosing to 1 hour after dosing. No food is allowed within 4 hours after dosing. During the study, subjects will receive standardized meals at approximately the same time each day.

SUMMARY:
This study is a single-site, open-label, single-cohort, single-dose study to assess the absorption, metabolism, and excretion profile of [14C] ABSK021 in healthy adult male subjects. The study plans to enroll 6 to 10 healthy male subjects to ensure at least 6 evaluable subjects.

DETAILED DESCRIPTION:
Subjects will be screened within 14 days before dose administration (D-14 to D-3), and will be admitted to the trial ward two days before dose administration (D-2).

On Day 1, subjects will receive a single oral dose of approximately 50 mg ABSK021 containing approximately 100 μCi of [14C] ABSK021 in the fasted state.

All excreted urine and feces samples and blood samples at specified time points during 0-504 hours after dosing will be collected. Random feces within 48 hours prior to dosing and random urine within 24 hours prior to dosing will be collected as blank samples (if there are multiple blank samples, the most recent blank sample before dosing will be selected for analysis).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who fully understand the content, procedures and possible adverse reactions before the study, and voluntarily sign the informed consent form, and can complete the study in accordance with the requirements in the protocol;
2. Healthy male subjects aged 18 to 45 years (including 18 and 45 years) at screening;
3. Weight ≥ 50 kg, body mass index (BMI) between 19 and 28 (including 19 and 28), BMI = weight (kg)/height (m) 2;
4. Subjects must have regular defecation in the past three months;
5. Male subjects of childbearing potential must agree to use effective contraceptive methods during the study and within 12 months after administration of study drug . Male subjects must agree to not donate sperm during this period.

Exclusion Criteria:

1. Abnormal and clinically significant complete physical examination, vital signs, digital rectal examination, laboratory tests (hematology, blood biochemistry, urinalysis, coagulation function, stool routine + occult blood, thyroid function, etc.), 12-lead electrocardiogram, chest X-ray (anteroposterior position), abdominal B ultrasound (hepatobiliary, pancreas, spleen and kidney);
2. Abnormal and clinically significant ophthalmic examination (slit lamp, intraocular pressure and fundus photography);
3. Tested positive for any one of the following: serum hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, treponema pallidum antibody (Syphilis) screening;
4. The baseline of heart rate corrected QT, QTcF interval prolongs > 450ms; family history of long QT syndrome (Note: QTc interval is corrected by Fridericia formula);
5. Creatinine clearance (CrCL) ≤ 60 mL/min, calculated using the Cockcroft-Gault formula ;
6. Subjects with a history of cardiovascular, respiratory, blood, liver, kidney, gastrointestinal, endocrine or nervous system diseases, for whom the absorption, metabolism or elimination of the drug are significantly affected, or for whom the investigator judges that the disease(s) may pose a risk when taking the test drug, interfere with the interpretation of the data, or affect the ability of the subjects to participate in the study;
7. Known or persistent mental disorders that may interfere with the subject's participation in the study, as judged by the investigator;
8. Known history of allergy to any drug or food;
9. Subjects who have participated in drug trials within 3 months before dosing.
10. Subjects who have participated in this study or any other study related to ABSK021, and have previously exposed to ABSK021;
11. Subjects who have used OATP1B1 inhibitors or strong CYP3A4 inhibitors or inducers (including grapefruit juice, grapefruit hybrids, pomegranates, carambola, grapefruit, Seville oranges and juice or other processed products) within 14 days prior to dosing;
12. Subjects with factors that significantly affect drug absorption, distribution, metabolism and excretion, such as inability to take the test drug orally, obvious nausea and vomiting and malabsorption; Subjects with history of gastric or intestinal surgery or resection (appendectomy and hernia repair surgery is allowed);
13. Subjects who are unwilling to comply with the dietary requirements/restrictions during the study. The specific dietary requirements are: (i) only eat the meals provided by the study sites during hospitalization, (ii) avoid consumption of OATP1B1 inhibitors or strong CYP3A4 inhibitors or inducers during this study;
14. Subject whose weekly alcohol consumption is greater than 14 units (1 unit of alcohol is equivalent to approximately 360 mL beer, 45 mL of spirits with 40% alcohol or 150 mL wine) within 3 months before dosing, or whose alcohol breath test result is ≥ 20 mg/dl;
15. Subjects who smoke more than 5 cigarettes per day (or an equivalent amount of tobacco or nicotine) within 3 months prior to dosing;
16. Subjects with overdose of methylxanthine/caffeine in the past 6 months as judged by the investigator (overdose is defined as more than 6 units of caffeine per day. 1 unit of caffeine is equivalent to 177 mL of coffee, 355 mL of tea, 355 mL of cola or 85 grams of chocolate);
17. Subjects with a history of bacterial, fungal, parasitic, viral (not including nasopharyngitis), mycobacterial infection within 45 days before dosing;
18. Known history of drug abuse or tested positive in drug abuse screening;
19. Subjects who have used or intend to use over-the-counter or prescription drugs, including herbal medicine, within 14 days prior to dosing and during the study;
20. Subjects who have donated plasma within 30 days before dosing or blood within 3 months before screening, or have experienced blood loss of > 400 mL;
21. A definite history of hemorrhoids; or perianal disease associated with regular hematochezia or ongoing bleeding, or habitual constipation/diarrhea;
22. Subjects who have been vaccinated within 2 months prior to dosing, or intend to be vaccinated throughout the study;
23. Subjects who have participated in the design or implementation of this project and their immediate family members (e.g., employees from Sponsor, CRO or research sites);
24. Subjects who need to work in a condition with long-term radioactive exposure, or who have experienced significant radioactive exposure (≥ 2 chest/abdominal CTs, or ≥ 3 other types of X-rays) within 1 year prior to the study, or who have participated in studies with radiopharmaceutical labelling;
25. Subjects with a history of needle sickness or blood sickness, who have difficulty or are intolerant to venipuncture;
26. Subjects with any other factors that may influence the participation in the study, which may affect the subject's compliance with the protocol, interfere with the interpretation of the study results, or expose the subject to risk, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion rate of radioactivity in excreta (urine, feces) and total radioactivity (urine and feces) | All excreted urine and feces samples at specified time points during 0-504 hours after dosing will be collected.
  To assess the routes and rates of elimination of ABSK021 and its metabolites after single oral administration of [14C]ABSK021 in healthy adult male subjects
Percentage of each metabolite in urine and feces relative to the administered dose (% administered dose), or percentage of metabolites in plasma relative to total exposure AUC (% AUC); | Conduct testing within 1 month after all subjects collect plasma, urine, and fecal samplesat all time points required by the protocol
  To determine the metabolism and elimination pathways of ABSK021 after single oral administration of [14C] ABSK021 in healthy adult male subjects, and identify major metabolites.All excreted urine and feces samples at specified time points during 0-504 hours after dosing will be collected.
Identification of major metabolites in plasma, urine, and fecal samples | Conduct testing within 1 month after all subjects collect plasma, urine, and fecal samplesat all time points required by the protocol
  To determine the metabolism and elimination pathways of ABSK021 after single oral administration of [14C] ABSK021 in healthy adult male subjects, and identify major metabolites.All excreted urine and feces and plasma samples at specified time points during 0-504 hours after dosing will be collected.
AUC 0-∞ | Conduct testing within 1 month after all subjects collect all samples at all time points required by the protocol
  To evaluate the pharmacokinetics of ABSK021 and its major metabolites in the urine of healthy adult male subjects after a single oral administration [14C] of ABSK021.
Tmax | Conduct testing within 1 month after all subjects collect PK samples at all time points required by the protocol
  To evaluate the pharmacokinetics of ABSK021 and its major metabolites in the fecal of healthy adult male subjects after a single oral administration [14C] of ABSK021

SECONDARY OUTCOMES:
Frequency, type and severity of adverse events/serious adverse events; changes in vital signs, 12-lead ECGs, laboratory tests, etc. | From signing the ICF until 22 days after the first dosing
  To assess the safety and tolerability of a single oral dose of approximately 50 mg with approximately 100 μCi [14C] ABSK021 in healthy adult male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Professor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of SOOCHOW UNIVERSITY, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No